CLINICAL TRIAL: NCT05244967
Title: Epidemiology of Sexually Transmitted Infections and Its iMpAcT on fEmale Infertility
Acronym: ESTIMATE
Status: Recruiting | Type: Observational
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Nadja Käding, PhD, University of Luebeck
Other Study IDs: 20-022
Record Dates: First submitted 2022-01-27; First posted 2022-02-17 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Sexually Transmitted Infection
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: vaginal swab — self-sampling, vaginal swab

SUMMARY:
A longitudinal study to investigate the prevalence of sexually transmitted infections among young women and determine the role of the female genital tract microbiome in fertility

ELIGIBILITY:
Inclusion Criteria:

* 18-22 years
* informed consent

Exclusion Criteria:

* pregnancy
* sterilization
* not capable of giving informed consent

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young women aged 18-22 years.
Sampling Method: Non-Probability Sample
Enrollment: 533 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
number of young women with STIs | at enrollment
  longitudinal analysis of STIs and the female genital tract microbiome
monitoring of STIs and their impact on infertility | through study completion, an average of 5 years
  obtain a better understanding for the emergence of infectious infertility and the impact on the pathogenicity

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Infektiologie und Mikrobiologie, Lübeck, Germany